CLINICAL TRIAL: NCT05405023
Title: Effects of Concentric Exercise With and Without Mulligan Wrist Mobilization on Pain, Grip Strength, Range of Motion and Function After Distal Radius Fracture.
Brief Title: Effects of Concentric Exercise With and Without Mulligan Wrist Mobilization After Distal Radius Fracture.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0128
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Distal Radius Fracture
Keywords: Disability; Range of Movement; Concentric exercises; Movement; Fracture
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentric exercises with wrist mobilization (Experimental): concentric exercise including wrist flexion, extension, and abduction, adduction, supination and pronation plus wrist mobilizations with movements
  Interventions: Other: Concentric exercises with wrist mobilization
- Concentric exercises without wrist mobilization (Active Comparator): concentric exercise including wrist flexion, extension, and abduction, adduction, supination and pronation
  Interventions: Other: Concentric exercises without wrist mobilization

INTERVENTIONS:
Other: Concentric exercises with wrist mobilization — Participants will receive concentric exercise including wrist flexion, extension, and abduction, adduction, supination and pronation plus wrist mobilizations with movements.
  Arms: Concentric exercises with wrist mobilization
Other: Concentric exercises without wrist mobilization — Participants will receive concentric exercises only.
  Arms: Concentric exercises without wrist mobilization

SUMMARY:
The distal end of the radius is defined as the area three centimeters proximal to the radio carpal joint, where the radius interfaces with the lunate and scaphoid bone of the wrist. A fracture of the distal radius is usually caused by falling on the outstretched arm. The majority of distal radial fractures are closed injuries in which the overlying skin remains intact. Pain, swelling, bruising, deformity and deformity in the forearm or wrist are common. In women, the incidence of distal radial fracture increases with age from 40 years. The objective of this study will be to determine the Effects of Concentric exercises with and without mulligan wrist mobilization on pain, grip strength, Range of motion and function after distal radius fracture.

This study will be a randomized controlled trial and will be conducted in District Head Quarter hospital sheikhupura. The study will be completed in time duration of six months after the approval of synopsis and convenience sampling technique will be used. 18 subjects will be divided in two groups. Group A will follow concentric exercises at wrist including flexion, extension, abduction, adduction, pronation, supination and wrist mobilizations with movements while group B will follow only wrist concentric exercises treatment. MWM based on Mulligan's Recommendation that the patient should not experience any pain. The Location and direction of the glide could be modified so that the MWM was pain free, as advocated in the Mulligan concept. This study will be of 4 weeks, 3 sessions per week. Data will be collected by all participants before 1st session after 6th session and at the end of 12th session by using NPRS, Hand Dynamometer, Goniometer and Patient Rated Wrist Evaluation score. Data will be analyzed by SPSS-25.

ELIGIBILITY:
Inclusion Criteria:

* Age: 35-70 years
* Subjects with at least 6 weeks of distal radius fracture
* Orthopedic surgeon advise

Exclusion Criteria:

* Neurological problem affecting upper limb
* Parkinson disease
* Subjects having polyarthritis, bleeding disorders, tumors, local infection, peripheral vascular disease
* Any contraindication to physiotherapy

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-05-27 (Estimated); Primary Completion 2022-11-27 (Estimated); Study Completion 2023-01-27 (Estimated)

PRIMARY OUTCOMES:
Wrist Pain | 4 weeks
  NPRS is anchored by terms describing pain severity extremes. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Grip Strength | 4 weeks
  Handheld dynamometers are used for measuring grip strength. They are available in manual and digital version so there is a need to know the reliability of manual hand-held dynamometer and digital hand-held for measuring grip strength. Excellent reliability is found for manual and digital handheld dynamometers
Range of motion | 4 weeks
  Goniometer is used to measure Range of motion. Hand-held pencil (HHP) and the plumb line goniometer (PLG) methods are used for measuring active forearm pronation and supination motions in individuals with and without injuries. The HHP and PLG are highly reliable methods for measuring functional forearm pronation and supination. Because plumb line goniometers are not commercially available and the instrumentation for the HHP method is readily accessible, clinicians should consider the latter as their method of choice for measuring functional forearm pronation and supination
Wrist Function | 4 weeks
  For evaluating function Patient Rated Wrist Evaluation (PRWE) score is used. High-quality evidence supports the use of PRWE/PRWHE as a reliable, valid, and structurally sound questionnaire to assess pain and disability in patients with various wrist and hand injuries. The PRWE/PRWHE has been translated into 21 languages. High-quality evidence supports very good structural and cross-cultural validity, internal consistency, test-retest reliability, measurement error, and hypothesis testing for construct validity against DASH in wrist and hand injuries. However, low-quality evidence supports acceptable responsiveness property

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, Phd*, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital Sheikhupura, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meena S, Sharma P, Sambharia AK, Dawar A. Fractures of distal radius: an overview. J Family Med Prim Care. 2014 Oct-Dec;3(4):325-32. doi: 10.4103/2249-4863.148101. PMID 25657938
- [Background] Quadlbauer S, Pezzei C, Jurkowitsch J, Rosenauer R, Kolmayr B, Keuchel T, Simon D, Beer T, Hausner T, Leixnering M. Rehabilitation after distal radius fractures: is there a need for immobilization and physiotherapy? Arch Orthop Trauma Surg. 2020 May;140(5):651-663. doi: 10.1007/s00402-020-03367-w. Epub 2020 Mar 19. PMID 32193679
- [Background] Gutierrez-Espinoza H, Rubio-Oyarzun D, Olguin-Huerta C, Gutierrez-Monclus R, Pinto-Concha S, Gana-Hervias G. Supervised physical therapy vs home exercise program for patients with distal radius fracture: A single-blind randomized clinical study. J Hand Ther. 2017 Jul-Sep;30(3):242-252. doi: 10.1016/j.jht.2017.02.001. Epub 2017 Mar 22. PMID 28342739
- [Background] Gutierrez-Espinoza H, Araya-Quintanilla F, Olguin-Huerta C, Valenzuela-Fuenzalida J, Gutierrez-Monclus R, Moncada-Ramirez V. Effectiveness of manual therapy in patients with distal radius fracture: a systematic review and meta-analysis. J Man Manip Ther. 2022 Feb;30(1):33-45. doi: 10.1080/10669817.2021.1992090. Epub 2021 Oct 20. PMID 34668847
- [Background] Coughlin T, Norrish AR, Scammell BE, Matthews PA, Nightingale J, Ollivere BJ. Infographic: Comparison of rehabilitation interventions in nonoperatively treated distal radius fractures: a randomized controlled trial of effectiveness. Bone Joint J. 2021 Jun;103-B(6):1031-1032. doi: 10.1302/0301-620X.103B6.BJJ-2021-0729. No abstract available. PMID 34058884
- [Background] Gutierrez-Espinoza H, Araya-Quintanilla F, Olguin-Huerta C, Gutierrez-Monclus R, Jorquera-Aguilera R, Mathoulin C. Effectiveness of early versus delayed motion in patients with distal radius fracture treated with volar locking plate: A systematic review and meta-analysis. Hand Surg Rehabil. 2021 Feb;40(1):6-16. doi: 10.1016/j.hansur.2020.10.007. Epub 2020 Nov 2. PMID 33144249
- [Background] Tomruk M, Gelecek N, Basci O, Ozkan MH. Effects of early manual therapy on functional outcomes after volar plating of distal radius fractures: A randomized controlled trial. Hand Surg Rehabil. 2020 May;39(3):178-185. doi: 10.1016/j.hansur.2019.12.002. Epub 2020 Feb 15. PMID 32070793
- [Background] Reid SA, Andersen JM, Vicenzino B. Adding mobilisation with movement to exercise and advice hastens the improvement in range, pain and function after non-operative cast immobilisation for distal radius fracture: a multicentre, randomised trial. J Physiother. 2020 Apr;66(2):105-112. doi: 10.1016/j.jphys.2020.03.010. Epub 2020 Apr 11. PMID 32291223
- [Background] Aguilera-Godoy A, Antunez-Riveros MA, Carrasco-Penna G, Nunez-Cortes R. A post-surgical rehabilitation program for women over 60 years old who underwent surgery in trauma and orthopedic hospital after distal radius fracture. J Bodyw Mov Ther. 2021 Oct;28:362-368. doi: 10.1016/j.jbmt.2021.07.042. Epub 2021 Aug 10. PMID 34776165
- [Background] Stathopoulos N, Dimitriadis Z, Koumantakis GA. Erratum to "Effectiveness of Mulligan's mobilization with movement techniques on pain and disability of peripheral joints: a systematic review with meta-analysis between 2008-2017" [Physiotherapy 105 (March (1)) (2019) 1-9]. Physiotherapy. 2020 Mar;106:219. doi: 10.1016/j.physio.2019.04.002. Epub 2019 Aug 30. No abstract available. PMID 31477334
- [Background] Shafiee E, MacDermid J, Farzad M, Karbalaei M. A systematic review and meta-analysis of Patient-Rated Wrist (and Hand) Evaluation (PRWE/PRWHE) measurement properties, translation, and/ or cross-cultural adaptation. Disabil Rehabil. 2022 Nov;44(22):6551-6565. doi: 10.1080/09638288.2021.1970250. Epub 2021 Sep 10. PMID 34505793